CLINICAL TRIAL: NCT04070742
Title: A 4-Day, Randomized, Controlled Study to Evaluate the Phototoxicity Potential of FMX-101, 4% in Healthy Volunteers
Brief Title: Dermal Phototoxicity Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX2016-06
Record Dates: First submitted 2019-08-08; First posted 2019-08-28 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMX-101 (Experimental)
  Interventions: Drug: FMX101

INTERVENTIONS:
Drug: FMX101

SUMMARY:
Dermal Safety study to determine the Phototoxicity Potential of FMX-101 4% in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers age 18 years or older
2. Has uniformly-colored skin on the lower thoracic area of the back which allowed discernment of erythema, and were Fitzpatrick Skin Types I, II, or III

Exclusion Criteria:

1. Has any visible disease at the application site which, in the opinion of the investigative personnel, would have interfered with the evaluation of the test site reaction
2. Are unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison between Test and Vehicle sites of the post-irradiation erythema severity at 96 hours post-application using a dermal response numerical equivalent score | 4 days